CLINICAL TRIAL: NCT02231541
Title: Effectiveness of Very Low Frequency Magnetic Fields in the Treatment of Fibromyalgia
Brief Title: Very Low Frequency Magnetic Fields in the Treatment of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, medical director, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3295/2014
Record Dates: First submitted 2014-08-08; First posted 2014-09-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2014-09

CONDITIONS: Fibromyalgia
Keywords: Fibromylgia; Magnetic Fields; Pain; Visual Analogue scale
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Very low frequency magnetic fields (Experimental): The very low frequency magnetic fields (ELF) are magnetic fields already use for orthopedics pathology that have shown to be able to repair, to reduce pain, inflammation and edema in the damaged tissues.
  Interventions: Device: Very Low Frequency Magnetic Fields
- Turned off very low frequency magnetic fields (Placebo Comparator): The very low frequency magnetic fields (ELF) are magnetic fields already use for orthopedics pathology that have shown to be able to repair, to reduce pain, inflammation and edema in the damaged tissues.
  Interventions: Device: Very Low Frequency Magnetic Fields

INTERVENTIONS:
Device: Very Low Frequency Magnetic Fields — The device is set to an analgesic program lasting about 30 minutes.
  Other Names: ELF
  Arms: Very low frequency magnetic fields
Device: Very Low Frequency Magnetic Fields — The device is turned off.
  Other Names: ELF
  Arms: Turned off very low frequency magnetic fields

SUMMARY:
The purpose of the study is to determine the effectiveness of treatment with very low frequency electromagnetic fields on the reduction of pain in patients with fibromylgia, disease presenting with widespread musculoskeletal pain usually associated with other symptoms such as stiffness, fatigue, sleep disturbances, depression, anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosed according to the criteria proposed by the American College of Rheumatology (ACR 2010)
* Subjects aged between 18 and 60 years

Exclusion Criteria:

* Pregnant patients
* Patients with pacemaker or other metal implants
* Systemic infectious disorders
* Neoplastic disorders
* Epilepsy
* Severe heart disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change of Visual Analogue Scale (VAS) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It is a scale for the assessment of pain and it's based on a ten point scale, where 0 means no pain and 10 the greatest pain ever both at rest and during movements.

SECONDARY OUTCOMES:
Change of Fibromylgia Impact Questionnaire (FIQ) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  The questionnaire assesses disability and symptoms. It is divided into ten sub-categories that assess the range of symptoms presented by the patient and the response to therapy and structured in twenty questions that assess disability in activities of daily living (ADL), the difficulties in practice, the feeling of general well-being, sleep, severity of symptoms, including pain, fatigue, depression, anxiety and rigidity. The questionnaire is self-administered disease-specific, and each item is based on a metric scale ranging from 0 (no disability) to 10 (maximum disability).
Change of Fibromylgia Assessment Status (FAS) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  The questionnaire assesses the response to therapy and the progression of the disease. Specifically it evaluates fatigue, sleep disorders and pain. The questionnaire is disease-specific, self-administered and is constituted by a "pain map", called Self-Assessment Pain Scale (SAPS) characterized by a metric scale from 0 to 3 and by two numerical scales for the assessment of fatigue and sleep quality, each characterized by a metric scale between 0 and 106.
Change of Health Assessment Questionnaire (HAQ) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  This questionnaire assesses disability. It is divided into eight domains that assess the dressing, eating, getting up, walking, hygiene, activities of achievement and activities of daily life. The questionnaire is self-administered and each item is based on a metric scale ranging from 0 (no disability) to 3 (maximum disability).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Principal Investigator — Umberto I Hospital, Sapienza University of Rome
Locations (1):
- Umberto I Hospital, Rome, Italy

REFERENCES:
- [Derived] Paolucci T, Piccinini G, Iosa M, Piermattei C, de Angelis S, Grasso MR, Zangrando F, Saraceni VM. Efficacy of extremely low-frequency magnetic field in fibromyalgia pain: A pilot study. J Rehabil Res Dev. 2016;53(6):1023-1034. doi: 10.1682/JRRD.2015.04.0061. PMID 28475205